CLINICAL TRIAL: NCT01841034
Title: Evaluation of a 6 Months Treatment of Conceptio (EA) on Sperm Data in Infertile Men With Oligoasthenozoospermia
Brief Title: Impact of an Antioxidant Alimentary Complement on Sperm Data
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 11-PP-13
Record Dates: First submitted 2011-09-26; First posted 2013-04-26 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Infertility
Keywords: Male
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Conceptio: Any patient receipt within the framework of the coverage(care) of an infertility in the pole ORG, whatever is the étiologie and the type of treatment proposing and presenting during at least two spermogrammes an oligospermie and\or an asthénospermie. The necessity of realizing 2 spermogrammes different to determine the pathological character of the values of a spermogramme takes into account the personal variability of the results.
  Interventions: Drug: Conceptio EA

INTERVENTIONS:
Drug: Conceptio EA — The patients are included during a consultation whether it is with a clinician or a biologist of the Center. It is suggested in routine in the service, to all the patients consulting for a problem of infertility and presenting pathological spermatic data, taking the food complement Conceptio. At the patients wishing to take this complement it will be suggested participating in this study. This complement is usually bought by the patient, within the framework of this study this one will be gracefully supplied. The follow-up of the patient will contain no examination and no anybody visit besides the usually realized follow-up.

SUMMARY:
Male infertility is a multifactorial disease process with a number of potential contributive causes. Considering the majority of male infertility cases are due to deficient sperm production of unknown origin, environmental and nutritional factors must be evaluated. The purpose of this study is to evaluate the effects of 6 months antioxidant dietary complement (Conceptio) on sperm parameters (sperm count, motility and DNA fragmentation) in infertile men with oligoasthenozoospermia.

ELIGIBILITY:
Inclusion Criteria:

* Number of sperm cells < 15M / mL and\or mobility < 40 %.
* Signature of a form of not opposition to the research.
* Membership in a social security system.

Exclusion Criteria:

* Number of sperm cells = 100M / mL.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient receipt within the framework of the care of an infertility in the pole ORG, whatever is the étiologie and the type of treatment proposing and presenting during at least two spermogrammes an oligospermie and\or an asthénospermie.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-05-30 (Actual); Primary Completion 2014-08-30 (Actual); Study Completion 2015-06-18 (Actual)

PRIMARY OUTCOMES:
Spermatic parameters (numeration and mobility spermatic) | At the inclusion and 6 months after the inclusion
  The spermatic parameters used within the framework of the spermogramme made in routine in the Laboratory of Biology of the Reproduction will be the numeration and the spermatic mobility from the very beginning.

SECONDARY OUTCOMES:
Rate of fragmentation of the DNA | At the inclusion and 6 months after the inclusion
  We shall consider the rate of fragmentation of the DNA determined according to the method of the TUNEL. This technique allows to estimate the rate of spermatozoides apoptose. It brings to light the fragmentation of the spermatic DNA in the course of process of cellular death.

CONTACTS AND LOCATIONS:
Overall Officials: ISNARD Véronique, PH, Principal Investigator — CHU de Nice - CECOS- Hôpital de l'Archet - 151 Route de saint-antoine de ginestière 06200 Nice
Locations (1):
- CHU de Nice - Hôpital de l'Archet, Nice, Alpes-Maritimes, France